CLINICAL TRIAL: NCT01430871
Title: Effects of Serotonin Excess on Bone in Carcinoid Syndrome
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Other Study IDs: STH15805
Record Dates: First submitted 2011-08-26; First posted 2011-09-08 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Carcinoid Syndrome
MeSH Terms: conditions — Serotonin Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 24 hour urine collections serum samples whole blood samples blood spot on cards
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Carcinoid syndrome: Patients: Men and women age 18 years or older with carcinoid syndrome attending the Sheffield neuro-endocrine tumour clinic
- Healthy Volunteers: Control group: Healthy men and women individually matched to the patients by gender, age, height and BMI

SUMMARY:
Serotonin has recently been identified as a major regulator of bone formation. Gut-derived serotonin inhibits bone formation, and early animal studies have shown that inhibition of gut-derived serotonin has anabolic effects on bone in ovariectomised rodents. This pathway has potential to be developed as a new anabolic treatment for osteoporosis in humans.

Carcinoid neuro-endocrine tumours produce very high levels of serotonin, and so it might be expected that patients with carcinoid disease would have reduced bone formation, low bone mass and fractures. However, this has not been apparent in clinical practice. There may be a discrepancy between rodent models and human disease. This study aims to identify whether patients with carcinoid disease have reduced bone mass, reduced bone formation or high fracture rates. The investigators will conduct a cross-sectional observational case-control study of patients with carcinoid disease in the Sheffield neuro-endocrine tumour clinic and gender-, age- and body mass index (BMI)-matched controls.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate
* Able to give informed consent
* Patient with carcinoid syndrome-active disease (untreated or receiving medical treatment)
* or
* Healthy volunteer who adequately matches a patient with carcinoid syndrome gender, age (±5 years), height (±5cm) and BMI(±3 kg/m2)

Exclusion Criteria:

* Curative surgery for carcinoid disease
* Body weight over 159 kg (weight limit for DXA measurement of BMD)
* Previous orthopaedic surgery or fractures which preclude imaging at all sites
* History of any long term immobilization (duration greater than three months)
* Fracture less than one year prior to recruitment
* Current pregnancy or trying to conceive
* Delivery of last child less than one year prior to recruitment
* Breast feeding less than one year prior to recruitment
* History of, or current conditions known to affect bone metabolism

  * Diagnosed skeletal disease or inflammatory arthritis
  * Chronic renal disease
  * Malabsorption syndromes
  * Other diagnosed endocrine disorders
  * Hypocalcemia or hypercalcemia
  * Diagnosed restrictive eating disorder
  * Diabetes mellitus
* Conditions or surgery which prevent the acquisition or analysis of DXA, VFA or HR-pQCT
* Use of medications or treatment known to affect bone metabolism
* Alcohol intake greater than 21 units per week

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women age 18 years or older with carcinoid syndrome attending the Sheffield neuro-endocrine tumour clinic Healthy men and women individually matched to the patients by gender, age, height and BMI
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2011-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Lumbar spine and total hip Bone Mineral Density BMD) measured by Dual-emission X-ray absorptiometry (DXA)

SECONDARY OUTCOMES:
Self-reported fracture history
Vertebral fracture assessment
Radius and tibia geometry and microarchitecture by HR-pQCT
Serum osteocalcin
Blood serotonin and 5HIAA
24h urine 5HIAA | 24 hours
Serum type 1 procollagen (N-terminal)(PINP)
Bone Alkaline Phosphatase (BAP)
Carboxy-terminal collagen crosslinks (CTX)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer S Walsh, PhD, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Academic Unit of Bone Metabolism (Sheffield), Sheffield, South Yorks, United Kingdom